CLINICAL TRIAL: NCT04860284
Title: The Efficacy and Safety of Hydroxychloroquine for the Treatment Of Non-Severe COVID-19 in Adults in Uganda: A Randomized Open Label Phase II Clinical Trial
Brief Title: Hydroxychloroquine for Treatment of Non-Severe COVID-19
Acronym: HONEST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAKRIF/DVCFA/016/20
Record Dates: First submitted 2021-04-23; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): Participants will receive 400mg of hydroxychloroquine tablets 12-hourly on day 1 and 200mg 12-hourly on day 2 to day 5 in addition to standard of care treatment for COVID-19
  Interventions: Drug: Hydroxychloroquine tablets
- Control arm (No Intervention): Participants will receive only standard of care treatment for COVID-19

INTERVENTIONS:
Drug: Hydroxychloroquine tablets — Hydroxychloroquine tablets 400mg given orally 12 hourly on day 1 and 200mg 12 hourly on day 2 to 5
  Other Names: HCQ
  Arms: Intervention arm

SUMMARY:
Currently there are no proven treatments for COVID-19 and current standard therapy is supportive care with oxygen supplementation and treatment of symptoms. Several re-purposed and new drugs have been investigated but none is conclusive for efficacy against COVID-19 .Both Hydroxychloroquine(HCQ) and Chloroquine(CQ) have demonstrated activity against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and have been investigated in small clinical trials with contradicting reports on their benefits or harm in treatment of COVID-19 .Several authors agree that the use of HCQ for treatment of COVID-19 needs to be assessed in large randomized controlled trials

DETAILED DESCRIPTION:
Currently there are no proven treatments for COVID-19 and current standard therapy is supportive care with oxygen supplementation and treatment of symptoms. Several re-purposed and new drugs have been investigated but none is conclusive for efficacy against COVID-19.These include the antimalarial drugs- chloroquine(CQ) and hydroxychloroquine(HCQ), antivirals such as remdesivir and favipiravir and antiretroviral combination therapies such as lopinavir/ritonavir. Although hydroxychloroquine and chloroquine are readily accessible in Uganda and could be explore for treatment of COVID-19,current data regarding their efficacy and safety is scanty.

It is necessary to determine whether HCQ can be useful for treatment of Ugandan patients with COVID-19 for the following reasons : Firstly, the Ugandan population expresses a high level of variability with a younger population with more than 50% under the age of 15 years. Secondly, the population with co-morbid conditions like diabetes mellitus ,hypertension and cardiovascular disease is significantly lower compared to higher income countries. Preliminary data from the first 52 COVID-19 patients in Uganda treated with HCQ demonstrated faster symptom resolution although this did not reach statistical significance. Lastly, HCQ has not been tested in mild-moderate disease where hospitalization is not necessary and we therefore do not know whether it can lead to faster viral clearance, slow disease progression and reduce time to symptom clearance. Our main aim will be to determine if hydroxychloroquine can lead to faster viral clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed positive Polymerase chain reaction(PCR) test for SARS COV-2
* Adults of ≥ 18 years
* Evidence of a personally signed and dated informed consent document indicating that the participant(or their legal representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Patients with contraindication to the use of hydroxychloroquine e.g. known allergy to hydroxychloroquine
* Patients enrolled in another interventional study which may interfere with study results
* Patients on medication that are known to have clinically significant interactions with the study drug e.g. digoxin, piperaquine, lumefantrine.
* Patients presenting with severe/critically ill COVID-19 (World Health Organization Ordinal scale for clinical improvement score of 5 or more)
* Patients with a fever( temperature ≥ 37.5 degrees centigrade) and a positive rapid diagnostic test (RDT) result for malaria
* Patients with corrected QT interval (QTc) prolongation of > 450ms for males and >470ms for females
* Pregnant or breastfeeding women
* Patients on chronic hydroxychloroquine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
SARS COV-2 viral clearance | From randomization to day 6
  Attaining a negative PCR- test result i.e. 100% viral clearance

SECONDARY OUTCOMES:
Clinical and laboratory adverse events | From randomization to day 6
  Grade 3 or 4 adverse events
Time to symptom clearance | Randomization to day 10
  Time from randomization to symptom clearance
Pharmacokinetic-pharmacodynamic model demonstrating drug concentration | Randomization to day 8
  Exposure-outcome relationship of hydroxychloroquine
Sero-reversion to negative antibody test | From randomization to day 90
  Antibody sero-reversion

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Byakika-Kibwika, PhD, Principal Investigator — Makerere University
Locations (1):
- Namboole COVID-19 treatment unit, Kampala, Uganda

REFERENCES:
- [Derived] Byakika-Kibwika P, Sekaggya-Wiltshire C, Semakula JR, Nakibuuka J, Musaazi J, Kayima J, Sendagire C, Meya D, Kirenga B, Nanzigu S, Kwizera A, Nakwagala F, Kisuule I, Wayengera M, Mwebesa HG, Kamya MR, Bazeyo W. Safety and efficacy of hydroxychloroquine for treatment of non-severe COVID-19 among adults in Uganda: a randomized open label phase II clinical trial. BMC Infect Dis. 2021 Dec 6;21(1):1218. doi: 10.1186/s12879-021-06897-9. PMID 34872511